CLINICAL TRIAL: NCT05511246
Title: Venous Ethanol for Ischemic Left Ventricular Tachycardia
Brief Title: Venous Ethanol for Ventricular Tachycardia
Acronym: VELVET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADM00021434
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy
Keywords: Ventricular tachycardia; Coronary veins; Ethanol; Ablation
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Ethanol; Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Endocardial radiofrequency ablation of ventricular tachycardia
  Interventions: Procedure: Catheter ablation
- Venous ethanol (Experimental): Endocardial radiofrequency ablation of ventricular tachycardia combined with venous ethanol ablation of the tachycardia substrate
  Interventions: Drug: Venous ethanol; Procedure: Catheter ablation

INTERVENTIONS:
Drug: Venous ethanol — Cannulation of coronary vein or veins in the VT substrate and balloon injection of ethanol
  Other Names: Alcohol
  Arms: Venous ethanol
Procedure: Catheter ablation — Endocardial catheter ablation of VT substrate

SUMMARY:
Comparative effectiveness randomized clinical trial, comparing endocardial radiofrequency ablation alone vs radiofrequency ablation combined with venous ethanol in patients with ischemic ventricular tachycardia -Venous Ethanol for Left Ventricular Ischemic Ventricular Tachycardia -VELVET clinical trial

DETAILED DESCRIPTION:
Patients with ventricular tachycardia (VT) in the context of ischemic heart disease suffer from significant morbidity and mortality. Catheter ablation can improve outcomes but has suboptimal ablation results. Ethanol ablation via epicardial veins can add significant therapeutic value to catheter ablation by increasing reach to intramural VT substrates. Investigators will randomize patients with ischemic VT to either endocardial catheter ablation alone, or combined with venous ethanol (VE) ablation of coronary veins located on the epicardial aspect of the VT substrates. A combined primary endpoint: VT recurrence, procedural complications, hospitalization for cardiac causes, and death, will be measured over a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages of 18 and 85 years and with a prior ICD implant
* Diagnosed with ischemic cardiomyopathy: Prior myocardial infarction (pathological Q waves or imaging evidence of regional myocardial akinesis/thinning in the absence of a non-ischemic cause)
* One of the following VT events (within last 6 months): a) ≥3 episodes of VT treated with anti-tachycardia pacing (ATP) or anti-arrhythmic drugs; b) ≥1 appropriate ICD shocks; c) ≥3 VT episodes within 24 hr; d) sustained VT below detection rate of the ICD documented by EKG/cardiac monitor
* Patients deemed candidates for RF ablation of VT
* Able and willing to comply with pre-, post-, and follow-up requirements
* Willing to sign the informed consent

Exclusion Criteria:

* Serum creatinine >1.5 mg/dL, or creatinine clearance <30 ml/min
* Left ventricular (LV) ejection fraction ≤10%
* Mobile LV thrombus on echocardiography
* Absence of vascular access to the LV
* Disease process likely to limit survival to <12 months
* New York Heart Association class IV heart failure
* Cardiac surgery within the past 2 months (unless VT was incessant),
* Acute coronary syndrome in the past 2 months (acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on EKG)
* Another reversible cause of VT (e.g. electrolyte abnormalities, drug-induced arrhythmia)
* Severe aortic stenosis or mitral regurgitation with a flail leaflet
* Pregnancy
* Unwilling or unable to provide informed consent
* Covid-19 positive testing within 14 days of randomization procedure
* Enrolled, or planning to get enrolled, in another research study during his/her participation on the Velvet trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2027-12-12 (Estimated); Study Completion 2028-12-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular tachycardia recurrence | 0-12 months
  Detection of VT on defibrillator
Hospitalization for cardiac causes | 0-12 months
Severe procedural complications | 0-12 months
  Severe procedural complications include bleeding requiring transfusion, stroke or systemic embolization, pericardial tamponade, myocardial infarction, and vascular complications requiring surgery, plus cardiogenic shock requiring unplanned mechanical support.
Death | 0-12 months

SECONDARY OUTCOMES:
Procedural time | During procedure
  Total procedure time (minutes)
Need for unplanned mechanical hemodynamic support | During procedure
  Unplanned use of intra-aortic balloon pump or ventricular assist device during procedure (Yes/No)
Repeat ablation procedures, including epicardial | 0-12 months
  Need for repeat procedure (Yes/No)
All-cause mortality | 0-12 months
Appropriate ICD therapies: antitachycardia pacing and ICD shocks | 0-12 months
  Presence of appropriate ICD therapies on interrogation
Inappropriate ICD therapies: antitachycardia pacing and ICD shocks | 0-12 months
  Presence of inappropriate ICD therapies on interrogation
Change in ICD therapies compared to 3-months pre-randomization | 0-12 months
  Comparison of number of therapies on ICD interrogation
Vt storm | 0-12 months
  More than 2 episodes of VT within a 24h period
Sustained VT below detection rate | 0-12 months
Change in left ventricular ejection fraction (percent) | Before and 3 months post-procedure
  Measured before and 3 months after procedure
Quality of life measurement using SF-32 questionnaire | 0-12 months
  Scores range from 0 - 100; Lower scores = more disability, higher scores = less disability
Hospital admission for cardiac causes (including heart failure exacerbation) | 0-12 months
  Hospitalization due to cardiac arrhythmia, heart failure exacerbation and other cardiac causes (yes/no)
Antiarrhtyhmic therapy | 0-12 months
  Number of antiarrhythmic drugs before and after ablation
Freedom from VT after repeat procedures | 0-12 months
  Recurrence of VT (yes/no) including patients that have multiple ablations
Cardiac transplant or left ventricular assist device implantation | 0-12 months
  As a measure of deterioration of cardiac status, requirement of transplant of ventricular assist device implant (yes/no) will be compared
Fluoroscopy time | During procedure
  Total time of fluoroscopy use (minutes)
Total contrast agent used | During procedure
  Amount of radiographic contrast used (cc)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Valderrabano, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No